CLINICAL TRIAL: NCT00091858
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Study of Darbepoetin Alfa for the Treatment of Anemia of Cancer
Brief Title: Study of Darbepoetin Alfa for the Treatment of Anemia of Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20010103; NCT00098696 (obsolete NCT alias)
Record Dates: First submitted 2004-09-17; First posted 2004-09-21 (Estimated); Last update posted 2013-05-08 (Estimated); Status verified 2013-05

CONDITIONS: Anemia; Cancer
Keywords: Cancer-related anemia
MeSH Terms: conditions — Anemia; Neoplasms | interventions — Darbepoetin alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Darbepoetin alfa 6.75 mcg/kg Q4W (Experimental)
  Interventions: Drug: Darbepoetin Alfa
- Placebo Q4W (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Darbepoetin Alfa — 6.75 mcg/kg Q4W
  Arms: Darbepoetin alfa 6.75 mcg/kg Q4W
Drug: Placebo — Placebo Q4W
  Arms: Placebo Q4W

SUMMARY:
The purpose of this study is to evaluate the efficacy of darbepoetin alfa versus placebo in reducing the occurrences of red blood cell transfusions in subjects with anemia of cancer who are not receiving chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* subjects with non-myeloid malignancies
* anemia due to cancer
* ECOG status 0 to 2
* greater than or equal to 4-month expectancy
* greater than or equal to 18 years and of legal age for informed consent
* screening hemoglobin concentration less than or equal to 11.0g/dL
* adequate serum folate and vitamin B12
* adequate renal and liver function
* written informed consent

Exclusion Criteria:

* subjects currently receiving or planned to receive cytotoxic chemotherapy or myelosuppressive radiotherapy during the study or within 4 weeks before randomization
* in complete remission, as determined by the investigator
* subjects who have other diagnoses not related to the cancer which cause anemia (eg. gastrointestinal bleeding, renal disease, etc)
* documented history of pure red cell aplasia
* Known history of seizure disorder
* cardiac condition: uncontrolled angina, congestive heart failure, known ejection fraction less than 40%, or uncontrolled cardiac arrhythmia
* uncontrolled hypertension
* clinically significant systemic infection or chronic inflammatory disease present at the time of randomization
* iron deficiency
* known positive test for HIV infection
* previously suspected of or confirmed to have neutralizing antibodies to rHuEPO or darbepoetin alfa
* received rHuEPO or darbepoetin alfa therapy within 4 weeks of randomization
* less than 30 days since receipt of any investigational drug or device that is not approved by the applicable regulatory authority
* pregnant or breast feeding
* subject of reproductive potential who is not using adequate contraceptive precautions
* known hypersensitivity to mammalian-derived product or any other ingredients in the investigational product
* previously randomized into this study
* concerns for subject's compliance with the protocol procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000
Dates: Start 2004-04; Primary Completion 2006-10 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Occurrences of red blood cell transfusion | from study day 29 (week 5) to week 17

SECONDARY OUTCOMES:
Incidence of first red blood cell transfusion | from week 5 (study day 29) to week 17 (study day 119)
Change in hemoglobin concentration measured | from baseline (study day 1) to EOTP
Adverse events and serious adverse events | throughout study for subjects who received at least 1 dose of investigational product
Survival | deaths on study and deaths in long-term follow-up period for subjects who received at least 1 dose of investigational product
Incidence, if any, of neutralizing antibody formation to investigational product | throughout study for subjects who received at least 1 dose of investigational product

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Smith RE Jr, Aapro MS, Ludwig H, Pinter T, Smakal M, Ciuleanu TE, Chen L, Lillie T, Glaspy JA. Darbepoetin alpha for the treatment of anemia in patients with active cancer not receiving chemotherapy or radiotherapy: results of a phase III, multicenter, randomized, double-blind, placebo-controlled study. J Clin Oncol. 2008 Mar 1;26(7):1040-50. doi: 10.1200/JCO.2007.14.2885. Epub 2008 Jan 28. PMID 18227526
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/20010103_CT_listing_final.pdf
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/20010103_Clin_trials_listing_final1.pdf
- See also: FDA-approved Drug Labeling — http://www.aranesp.com/